CLINICAL TRIAL: NCT01942902
Title: A Comparative Study to Evaluate the Accuracy and Safety of the GlySure Continuous Intravascular Glucose Monitoring System Versus Intermittent Blood Glucose Monitoring Using the Yellow Springs Blood Glucose Analyser for Conformité Européenne (CE) Marking Purposes in a Total of Thirty Patients Admitted to The Surgical Intensive Care Unit (SICU)
Brief Title: A Comparative Study to Evaluate the Accuracy and Safety of the GlySure Continuous Intravascular Glucose Monitoring System Versus Intermittent Blood Glucose Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlySure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013.01.CE
Record Dates: First submitted 2013-08-15; First posted 2013-09-16 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Continuous Glucose Measurement
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Continuous Glucose Monitoring System (Experimental)
  Interventions: Device: Continuous Glucose Monitoring System

INTERVENTIONS:
Device: Continuous Glucose Monitoring System
  Other Names: Glysure

SUMMARY:
The purpose of this study is to evaluate the system performance of the GlySure Continuous Glucose Monitoring (CGM) system in patients admitted to the Surgical Intensive Care Unit.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or legal representative MUST be willing to sign an informed consent document
2. Male and female aged 18 years and above
3. Require Central Venous Catheter (CVC) into the right internal Jugular vein as part of disease management and treatment
4. Expected to remain in the Surgical Intensive Care Unit (SICU) for at least 30 hours and up to 7 days-

Exclusion Criteria:

1. Patient or legal representative unable to provide written informed consent
2. Patient who is pregnant
3. Patient who is currently being administered Mannitol
4. Patient with history of Pulmonary Embolism (PE)
5. Patient with history of thrombosis
6. Patient with known hyper-coagulation
7. Patient with known history of heparin hypersensitivity
8. Patient with history of heparin induced thrombocytopenia
9. Participation in a clinical study involving an unlicensed pharmaceutical product and/or device within the 3 months prior to enrolment in this study
10. Patient with known hypersensitivity/allergy to adhesive I.V. dressings such as 3M Tegaderm film
11. Patient likely to require an MRI scan during their stay in the SICU
12. Patients likely to require treatment with Mannitol during time in the SICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Accuracy of the CGM system as compared with the Yellow Springs Instrument (YSI) blood sample analysis results | For at least 30 hours and up to 7 days
  The study is designed to evaluate the comparative accuracy between measured blood glucose results obtained from the GlySure Continuous Glucose Monitoring System (CGM) and the YSI, and to determine if any condition or treatment affects the sensor's measured values.
Number of participants experiencing Serious Adverse Events (SAEs) causally related to the devices | For at least 30 hours and up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Prasad, MD, Principal Investigator — Care Hospital
Locations (2):
- India (2):
  - Star Hospital, Banjara Hills, Hyderabad
  - Care Hospital, Nampally, Hyderabad